CLINICAL TRIAL: NCT05387928
Title: A Phase 1 Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of KL340399 Injection in Patients With Advanced Solid Tumors
Brief Title: A Study of KL340399 in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sichuan Kelun-Biotech Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Sichuan Kelun Pharmaceutical Research Institute Co., Ltd. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KL296-I-01
Record Dates: First submitted 2022-05-19; First posted 2022-05-24 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dose Escalation (Experimental): KL340399 weekly on Days 1, 8 and 15 on repeated 21-day cycles in escalating doses.
  Interventions: Drug: KL340399 injection

INTERVENTIONS:
Drug: KL340399 injection — KL340399 injection is a STING-activating. The strength of KL340399 is 0.2 mg/vial，0.2 mg/vial.

SUMMARY:
This is a single center, open-label, dose increasing study to evaluate the safety, tolerability, pharmacokinetic(PK) profile, and antitumor efficacy of KL340399 injection in patients with advanced solid tumors.

DETAILED DESCRIPTION:
This is a single center, open-label, dose increasing study to evaluate the safety, tolerability, pharmacokinetic(PK) profile, and antitumor efficacy of KL340399 injection in patients with advanced solid tumors.The dose increasing method of "BLRM" is used to explore the safety, tolerance and determine the maximum tolerated dose(MTD).

ELIGIBILITY:
Inclusion Criteria:

1. Patient is at least ≥18 years of age (male or female);
2. Patients with histologically and/or cytologically confirmed advanced solid tumors who have failed standard of care, or who have no available standard of care regimen, or who are unqualified for standard of care. Presence of at least one measurable lesion based on Response Evaluation Criteria in Solid Tumors (RECIST) v1.1;
3. Eastern Cooperative Oncology Group (ECOG) score of 0 or 1, estimated survival ≥ 3 months;
4. Adequate organ and bone marrow function (no blood components and cytokines are allowed within 14 days prior to the first dose) ;
5. More than 4 weeks from the last radiotherapy, chemotherapy, surgery, hormone treatment, target therapy, and toxicity from previous antitumor therapy returned to baseline or CTCAE≤ grade 1;
6. Patients of childbearing potential (male or female) must use effective medical contraception during the study and for 3 months after the end of dosing;
7. Patients voluntarily participate in the study, sign the ICF, and will be able to comply with the protocol-specified visits and relevant procedures.

Exclusion Criteria:

1. Known history of severe allergies, or allergy to any component of KL340399;
2. Received any previous therapy of STING-activating, or received any immunostimulant therapy within 28 days；
3. Have other malignancies within 5 years;
4. Concomitant or known metastases to brain or central nervous system;
5. Active autoimmune disease;
6. History of major cardiovascular diseases;
7. Uncontrolled systemic diseases；
8. Known of coagulation disorders, hemorrhagic disease;
9. Confirmed serious lung disease or lung disease;
10. Subjects with third space fluid that can not be controled by drainage or other methods;
11. Known active infection;
12. Known HIV, active hepatitis B/C virus;
13. Pregnant or lactating women;
14. Received immunotherapy and had immune related adverse reactions ≥ grade 3;
15. Have received stem cell transplantation or organ transplantation;
16. Receive any live or attenuated live vaccine within 4 weeks;
17. History of serious dementia, altered mental status, or any psychiatric disorder;
18. Evidence of alcohol or drug abuse;
19. Participated in any other clinical trials and received treatment within 4 weeks;
20. Have other factors based on which the investigator considers that the subjects are not appropriate to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2022-06-07 (Actual); Primary Completion 2025-04-02 (Actual); Study Completion 2025-04-02 (Actual)

PRIMARY OUTCOMES:
Number of subjects achieving Dose-limiting toxicity (DLT) | From data of initial dose until up to 21 days for treatment
  DLT is defined as an adverse event (AE) that meets protocol defined DLT criteria during cycle 1 and is at least possibly related to study drug.
Maximum Tolerated Dose (MTD) | From data of initial dose until up to 21 days for treatment
  The maximum tolerated dose (MTD) is refers to the highest dose at which the patient's DLT incidence exceeding 33% during the first cycle.
Recommended Phase 2 Dose (RP2D) | Up to 24 months
  The recommended phase 2 dose (RP2D) will be based on a consideration of the totality of data including but not limited to safety data (including DLTs), PK, PD and preliminary efficacy, as available.
Incidence of Adverse Events [Safety and Tolerability] | Up to 24 months
  Incidence of adverse events of KL340399 as a monotherapy as determined by patient reporting, clinical laboratory test changes from baseline, and clinically significant changes in physical examination data.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Up to 24 months
  The sum of the number of cases with Complete Response (CR) and Partial Response (PR) in all treated tumor patients (CR + PR) divided by the total number of cases.
Progression Free Survival (PFS) | Up to 24 months
  PFS: Time from start of treatment to progression of disease (PD) or death, whichever occurs first, in patients with tumors.
Duration of Response (DOR) | Up to 24 months
  DOR: Time from the start of the first assessment of CR or PR in tumor patients to PD or death due to any reason.
Overall Survival (OS) | Up to 24 months
  OS: Time from start of treatment to death due to any reason.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Guo, Dr., Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China